CLINICAL TRIAL: NCT02131363
Title: A Clinical Investigation to Evaluate the Safety and Performance of a Treatment Kit for Ingrowing Toenail
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reckitt Benckiser Healthcare (UK) Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPD21402
Record Dates: First submitted 2014-05-02; First posted 2014-05-06 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2014-09

CONDITIONS: Onychomycosis of Toenails

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ingrowing Toenail Treatment Kit (Experimental): Ingrowing Toenail Treatment Kit consists of 3 components:
  1. Toe nail clip: one clip to be applied each week, for 6 weeks.
  2. Aerosol spray: to be applied up to 5 times a day, no more than one spray per hour.
  3. Nail adhesive: used to attach the clip to the nail.
  Interventions: Device: Ingrowing Toenail Treatment Kit

INTERVENTIONS:
Device: Ingrowing Toenail Treatment Kit — detailed in arm description

SUMMARY:
This purpose of this study is to evaluate the safety and performance of a treatment kit for ingrowing toenail, primarily by determining the number of subjects who show a reduction in the severity of their ingrowing toenail.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with one great ingrowing toenail that is rated as either "slightly ingrowing", "somewhat ingrowing" or "very ingrowing" on the Investigators Ingrowing Toenail Severity Scale.
* Subjects whose worst pain experienced in the week preceding inclusion, is rated at least 3 on the 10 point Subject Pain Intensity Scale.
* Subjects whose affected toenail has a minimum of 2mm distal edge and a minimum nail width of at least 16mm.

Exclusion Criteria:

* Subjects with any other toenail pathology (including pincer and spicule toenail) that would compromise the fitting of the toenail clip, or its use.
* Subjects suspected to be immunocompromised.
* Subjects who suffer from impaired feeling in the feet due to diabetes, peripheral vascular disease or neuropathy.
* Subjects with any cutaneous pathology or cuts/abrasions which, in the opinion of the investigator, could compromise safety or affect the outcome of the clinical investigation (for example, interfere with assessments).
* Subjects with known sensitivity/allergies to any component of the investigational device.
* Significant current or past medical history of hepatic, renal, cardiac, pulmonary, digestive, haematological, neurological, locomotor or psychiatric disease, which, in the opinion of the Investigator, would compromise the safety of the subject or affect the outcome of the clinical investigation (as determined from self-reported medical history questionnaire).
* Use of concomitant medication likely to affect the response to the investigational device or confuse the results of the clinical investigation. Regular pain relief is not permitted and subjects must not take any analgesics in the 24 hours preceding any clinic visit.
* Female subjects of childbearing potential who, for the duration of the study, are either unwilling or unable to take adequate contraceptive precautions or are unwilling to be sexually abstinent.
* Pregnancy or lactating mother.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-08; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects who demonstrate a reduction in the severity of their ingrowing toenail | At Day 42 from Day 0
  This will be assessed by the Investigator, using the Investigator Ingrowing Toenail Severity Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- CPS Research Ltd., Glasgow, Scotland, United Kingdom